CLINICAL TRIAL: NCT04203121
Title: The Safety and Scientific Validity of Low-dose Whole Brain Radiotherapy on Brain Amyloidosis During the Treatment of Mild or Moderate Alzheimer's Disease.
Brief Title: The Safety and Scientific Validity of Low-dose Whole Brain Radiotherapy in Alzheimer's Disease.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyung Hee University Hospital at Gangdong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KHNMC 2018-09-022-003
Record Dates: First submitted 2019-11-21; First posted 2019-12-18 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2019-09

CONDITIONS: Alzheimer Disease
Keywords: radiotherapy
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: arm 1 :subjects 1-5 - 9Gy in 5 daily fractions
  arm 2 :subjects 6-10 - 5.4Gy in 3 daily fractions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arm1 (Experimental): An initial 5 patients will be enrolled in the first treatment scheme and will be followed for 6 months after completion of treatment to assess safety and any toxicity events associated with treatment.
  subjects 1-5 : 9 Gy in 5 fractions of 1.8 Gy on 5 consecutive days
  Interventions: Radiation: low dose whole brain radiation to treat Alzheimer disease
- arm2 (Experimental): Subjects in this arm will be enrolled in the second treatment scheme and will be followed for 6 months after completion of treatment to assess safety and any toxicity events associated with treatment.
  subjects 6-10 : 5.4 Gy in 3 fractions of 1.8 Gy on 3 consecutive days
  Interventions: Radiation: low dose whole brain radiation to treat Alzheimer disease

INTERVENTIONS:
Radiation: low dose whole brain radiation to treat Alzheimer disease — subjects 1-5 : 9Gy in 5 daily fractions
  subjects 6-10 : 5.4Gy in 3 daily fractions

SUMMARY:
Alzheimer's disease is the most frequent neurocognitive disorder associated with dementia, with a constantly increasing prevalence associated with an aging population. Amyloid deposition is considered as the first molecular event on the onset of Alzheimer's disease. It has already been demonstrated that low-dose radiotherapy is capable of reducing Alzheimer's disease-associated amyloid-β plaques and improving cognitive function in an animal model. In human, low-dose radiotherapy has demonstrated effectiveness in reducing bronchial amyloidosis.

The present study aims to conduct research by including 10 patients with a diagnosis of mild or moderately severe Alzheimer's disease and with evidence of amyloid pathology. Furthermore, the aim is to demonstrate the effectiveness of low-dose radiotherapy in reducing amyloid deposits in the human brain using molecular imaging (Flutemetamol(18F) PET) along with treatment of the specific target.

DETAILED DESCRIPTION:
The investigators decided to use fractionated whole brain radiation doses of 1.8 Gy x 5 and 1.8 Gy x 3. Subjects will be followed with neurocognitive testing at 6 months post radiotherapy.

subjects 1-5 - 9Gy in 5 daily fractions

subjects 6-10 - 5.4Gy in 3 daily fractions

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of mild or moderate Alzheimer's disease.
* Amyloid PET scan positivity.
* Korean Mini-Mental State Examination score ≥10 and ≤24.
* Clinical dementia rating scale 0.5, 1 or 2.
* Ability to undergo neurocognitive assessment at baseline visit, alone or accomparined by a caregiver.
* Ability to understand the clinical trial and give an informed consent

Exclusion Criteria:

* previous therapeutic whole brain irradiation
* Evidence of seizure activity
* Evidence of active dermatological skin disease of the scalp.
* History of malignant tumors.
* Pregnant or breastfeeding.
* If the researcher determines that participation in this study is inadequate because of other findings that are considered clinically important.

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate low-dose whole brain radiotherapy in subjects with early Alzheimer's dementia using neurocognitive testing methods | 6 months after the first visit.
  verification of radiation therapy effect through GDS test

SECONDARY OUTCOMES:
change in brain amlyoid deposits | 6 months after the first visit
  The change in SUV of the frontal, parietal, extramedullary, pre-wedge, and posterior fasciocutaneous flutemetamol (18F) PET is considered to be an effective response if the change in SUV is more than 5%.

CONTACTS AND LOCATIONS:
Locations (1):
- Kyung Hee University Hospital at Gangdong, Seoul, South Korea